CLINICAL TRIAL: NCT04247178
Title: NIPPA: Non-Invasive Haemoglobin Measurement to Identify Preoperative Anaemia in Patients Scheduled for Elective Orthopaedic Surgery, a Single-centred Prospective Cohort Study.
Brief Title: Non-invasive Identification of Preoperative Anaemia
Acronym: NIPPA
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC19147
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Patients undergoing elective orthopaedic surgery
- Healthy Volunteers

SUMMARY:
Approximately 20% of patients undergoing elective orthopaedic surgery are anaemic. When not identified and treated before surgery, this can lead to requiring blood transfusions, which brings additional expenses, time and inconvenience to the patient.It is recommended that preoperative assessment involves investigation and where possible, treatment of anaemia.

The timescale between assessment and surgery makes it difficult to comply with guidelines without postponing surgery.

This study will investigate adult patients scheduled for elective orthopaedic surgery, where a full blood count is to be taken as part of routine care. A paired non-invasive reading of their blood will be taken. It will be conducted at The Royal Infirmary, Edinburgh. This device is not in use within the department currently but has been given free of charge for the study. There are no restrictions placed on the device except that it is not accurate for measuring haemoglobin <8g.dL. Participant care will only be determined by results from the laboratory assay as per routine care, not the noninvasive device.

The device is CE marked for haemoglobin determination. Masimo (manufacturer) have released results in the accuracy of their monitor but with very little other information, for example, study population or precision. This study aims to answer how accurate and precise non-invasive measurements are in patients scheduled for orthopaedic surgery (there are no studies with these results) and whether anaemia can be identified earlier in the patient pathway i.e. an anaemia screen at time of surgical listing, therefore leaving ample time for treatment and optimisation of care.

The data from the study will not be shared with Masimo. There is ongoing work towards introducing and piloting a new pre-operative triage system where optimisable conditions e.g. anaemia are identified at the time of listing. This study would aid this work.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* aged between 16-80 years old
* scheduled for elective orthopaedic surgery
* a full blood count (FBC) is to be taken as part of routine care

Inclusion Criteria for healthy volunteers cohort:

* able to provide informed consent
* aged between 16-80 years old

Exclusion Criteria:

* Patients with haemoglobin disorders
* Raynaud's disease (or any other condition affecting the blood supply to the digits).

Exclusion Criteria for healthy volunteers cohort:

* Patients with haemoglobin disorders
* Raynaud's disease (or any other condition affecting the blood supply to the digits).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for elective orthopaedic surgery.
  Healthy volunteers will be recruited from The Department of Anaesthetics.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
The accuracy of the non-invasive device | January to March 2020
  assessed by calculating the agreement between the results obtained from the gold standard laboratory assay and the non-invasive device

SECONDARY OUTCOMES:
Correlation of the non-invasive device to the gold standard | January to March 2020
  Intraclass correlation coefficient
Correlation of the non-invasive device to the gold standard | January to March 2020
  Interclass correlation coefficient
Predictive value of the non-invasive device | January to March 2020
  sensitivity
Predictive value of the non-invasive device | January to March 2020
  specificity
Predictive value of the non-invasive device | January to March 2020
  positive predictive value
Predictive value of the non-invasive device | January to March 2020
  negative predictive value
Factors independently associated with bias | January to March 2020
  age in years
Factors independently associated with bias | January to March 2020
  sex (male or female)
Factors independently associated with bias | January to March 2020
  perfusion index measured by noninvasive device
Factors independently associated with bias | January to March 2020
  pleth variability index measured by noninvasive device low signal quality
Factors independently associated with bias | January to March 2020
  heart rate measured by noninvasive device low signal quality
Factors independently associated with bias | January to March 2020
  SpO2 (peripheral oxygen saturation) measured by noninvasive device low signal quality
Factors independently associated with bias | January to March 2020
  low signal quality measured by noninvasive device low signal quality

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, The City of Edinburgh, United Kingdom